CLINICAL TRIAL: NCT04110639
Title: Intraoperative Monitoring of Femoral Head Perfusion in Femoral Neck Fractures
Brief Title: Intraoperative Monitoring of Femoral Head Perfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Children's Healthcare of Atlanta (Other)
Collaborators: Geogia Trauma Foundation (Unknown)
Responsible Party: Principal Investigator, TIm Schrader, MD, Principal Investigator, Children's Healthcare of Atlanta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-148
Record Dates: First submitted 2019-09-15; First posted 2019-10-01 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Monitoring, Physiologic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Validation Group (Active Comparator): A validation group of 10 patients with minimally displaced femoral neck fractures (Garden 1) which will be pinned in situ without manipulation
  Interventions: Other: Standard of Care
- Study Group (Experimental): A study group of 20 patients with displaced femoral neck fracture patients (Garden 2-4) treated with open or closed reduction and internal fixation
  Interventions: Device: Intracranial pressure (ICP) monitor

INTERVENTIONS:
Device: Intracranial pressure (ICP) monitor — The investigators' hypothesis is that by utilizing an intracranial pressure (ICP) monitor to detect the presence or absence of waveforms in the femoral head, investigators could reliably assess the perfusion levels within the femoral head and possibly reduce the incidence of osteonecrosis.
  Arms: Study Group
Other: Standard of Care — 10 patients with minimally displaced femoral neck fractures (Garden 1) which will be pinned in situ without manipulation
  Arms: Validation Group

SUMMARY:
An ICP monitor will be used to record blood flow/perfusion of the femoral head following fixation of femoral neck fractures. FDA approved device but not for this use.

DETAILED DESCRIPTION:
Hip fractures are a common entity in the realm of orthopedic trauma care and make up about 20% of the average workload of a trauma center. The lifetime risk of sustaining a hip fracture is significant; in women the range is 40-50% and among men it is 13-22%. Among all hip fractures, intracapsular femoral neck fractures (FNF) account for approximately 50% and are a significant undertaking for both the patient and treating physician. As the average age of the general population increases, the incidence of FNF in the worldwide population is likewise expected to rise (1.66 million observed in 1990 and 6.26 million projected 2050) with profound societal and economic impact.1

Operative indications and the methodology of surgical intervention in cases of femoral neck fractures are well established. Generally speaking, treatment options can be divided in two groups: reduction with internal fixation or arthroplasty. This treatment decision depends on patient factors and fracture characteristics. Within the realm of internal fixation, advances in the quality of modern implants have yielded largely good surgical outcomes. However, internal fixation of femoral neck fractures is not without complications. Osteonecrosis of the femoral head (ONFH) and nonunion are the major causes of morbidity and economic burden.2 The rate of ONFH in a recent meta-analysis was 0-22% (mean 6.9%) with a trend towards higher rates in women, patients less than 60 years of age, and those treated with cannulated screw fixation.1,3,4 Identifying measures to minimize the risk of osteonecrosis and nonunion would be beneficial to patient outcomes. Prior studies have noted correlations between residual displacement of the femoral head or varus malreduction with fixation failure (13-fold increase).1,5 In both cases, it is suspected that failure to restore normal anatomy of the femoral head and neck compromises the biomechanical alignment of the hip, and most importantly, its blood flow.

To date, there has not been a well-described intra-operative method to assess femoral head perfusion in adults, or to correlate these finding with late complications such as osteonecrosis. The diagnosis of osteonecrosis is typically made late in the patient's post-operative course when it becomes apparent on radiographs. Some investigators have studied the utility of select imaging studies at predicting femoral head perfusion and found single photon-emission computerized tomography (CT) to be accurate, but not easily available in all centers.6 MRI is felt to be superior to radiographs for early detection, but still not reliable in the first few weeks after injury.7 While the use of post-operative MRI and CT to elucidate femoral head perfusion has been investigated, neither can provide a real-time, intra-operative, measure of blood flow to the femoral head. If a real-time perfusion assessment tool was available, surgeons could determine the necessity for, and adequacy of, intraoperative reduction. Lack of perfusion could alter a surgeon's operative plan and might prompt an attempt at improving the reduction or a change in surgical management.

The purpose of this prospective study is to establish an intra-operative technique to monitor femoral head blood flow in patients with femoral neck fractures. The investigators' hypothesis is that by utilizing an intracranial pressure (ICP) monitor to detect the presence or absence of waveforms in the femoral head, investigators could reliably assess the perfusion levels within the femoral head and possibly reduce the incidence of osteonecrosis. Primary outcomes will be osteonecrosis and fracture union. The implications of this study may lead to changes in post-operative management, the intra-operative surgical plan if little to no epiphyseal perfusion is present and potentially new treatments for FNF patients to avoid the dreaded complication of osteonecrosis.

The intracranial pressure monitor will be utilized during the standard operative fixation of displaced and non-displaced FNF patients. This will allow a real-time assessment of femoral head perfusion pressure following reduction and fixation of these fractures. Correlations will be made to patients' blood pressure, demographic data, and injury characteristics. The monitor uses a sterile transducer that contains a pressure-monitoring catheter. This produces an artifact free, high fidelity waveform tracing without the need for a "fluid-filled" system. In the proposed application, the monitor would quantify perfusion pressure in the femoral head rather than cerebral tissue pressure. Following the investigators' protocol, the ICP monitor will be inserted through the cannulated screw used for fracture fixation and then removed after the measurement has been recorded.

Dr. Tim Schrader, the principal investigator, currently utilizes this ICP monitor as standard of care for all patients being treated for unstable slipped capital femoral epiphysis, a pediatric condition of the hip that similarly has an associated risk of osteonecrosis. He has demonstrated that the presence of femoral head perfusion as detected by a waveform on intra-osseous placed ICP monitor has been associated with the absence of osteonecrosis post-operatively.8

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Ages 1 to 18 years
* Acute femoral neck fracture
* Consent to enrollment

Exclusion Criteria:

* Hip fractures other than femoral neck fractures
* Femoral neck fractures treated with arthroplasty
* Absence of a consenting parent/guardian or parent/guardian unwilling to consent to participation
* Loss to follow-up

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Femoral Head Perfusion Monitoring | During surgery
  Establish an intra-operative technique to monitor femoral head blood flow in patients with femoral neck fractures.

SECONDARY OUTCOMES:
Reduce Osteonecrosis | Post-op: One Year after surgery
  By utilizing an intracranial pressure (ICP) monitor to detect the presence or absence of waveforms in the femoral head, investigators could reliably assess the perfusion levels within the femoral head and possibly reduce the incidence of osteonecrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Dedrick DK, Mackenzie JR, Burney RE. Complications of femoral neck fracture in young adults. J Trauma. 1986 Oct;26(10):932-7. doi: 10.1097/00005373-198610000-00013. PMID 3773004
- [Background] Maurer SG, Wright KE, Kummer FJ, Zuckerman JD, Koval KJ. Two or three screws for fixation of femoral neck fractures? Am J Orthop (Belle Mead NJ). 2003 Sep;32(9):438-42. PMID 14560825
- [Background] Min BW, Kim SJ. Avascular necrosis of the femoral head after osteosynthesis of femoral neck fracture. Orthopedics. 2011 May 18;34(5):349. doi: 10.3928/01477447-20110317-13. PMID 21598895
- [Background] Wang C, Xu GJ, Han Z, Jiang X, Zhang CB, Dong Q, Ma JX, Ma XL. Correlation Between Residual Displacement and Osteonecrosis of the Femoral Head Following Cannulated Screw Fixation of Femoral Neck Fractures. Medicine (Baltimore). 2015 Nov;94(47):e2139. doi: 10.1097/MD.0000000000002139. PMID 26632739
- [Background] Stromqvist B, Brismar J, Hansson LI, Palmer J. Technetium-99m-methylenediphosphonate scintimetry after femoral neck fracture. A three-year follow-up study. Clin Orthop Relat Res. 1984 Jan-Feb;(182):177-89. PMID 6229381
- [Background] Speer KP, Spritzer CE, Harrelson JM, Nunley JA. Magnetic resonance imaging of the femoral head after acute intracapsular fracture of the femoral neck. J Bone Joint Surg Am. 1990 Jan;72(1):98-103. PMID 2295679
- [Background] Schrader T, Jones CR, Kaufman AM, Herzog MM. Intraoperative Monitoring of Epiphyseal Perfusion in Slipped Capital Femoral Epiphysis. J Bone Joint Surg Am. 2016 Jun 15;98(12):1030-40. doi: 10.2106/JBJS.15.01002. PMID 27307364
- [Background] Keating, John. Rockwood and Green Chapter 49 - Femoral Neck Fractures p.2031-2070. Wolters Kluwer Health 2015. Philadelphia, PA.